CLINICAL TRIAL: NCT04719312
Title: Evaluation of Modification of the Transconjunctival Approach in Open Reduction of Zygomatic Maxillary Complex Fracture
Brief Title: Y Transconjunctival Approach in Open Reduction of Zygomatic Maxillary Complex Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y transconjunctival approach
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Zygomatic Fractures
MeSH Terms: conditions — Zygomatic Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- transconjunctival Y modification (Experimental)
  Interventions: Procedure: Y modification of transconjunctival approach

INTERVENTIONS:
Procedure: Y modification of transconjunctival approach — Section of the orbital septum is done at the Arcus Marginalis and subperiosteal dissection done to expose the infraorbital rim and orbital floor.
  Subsequently, canthotomy of the superficial limb of the lateral canthal ligament is performed and subperiosteal dissection is carried out to expose the fracture at the frontozygomatic region.
  The cutaneous Y will transform into a box when retracting its corners, increasing the working area and allowing access of the frontozygomatic (FZ) suture, lateral orbital wall, body of the zygoma, infraorbital rim, and floor of the orbit with a single approach.
  A small upper vestibular incision is placed to expose the fracture at the zygomatic buttress. Reduction and fixation of fractures in a regular fashion are accomplished.

SUMMARY:
this study was made on fifteen patients who will undergo fracture repair of the zygomaticomaxillary complex.

Postoperative patient evaluation performed with specific attention paid towards, accessibility the exposure duration(time from incision till exposure of the field), esthetic appearance, post-operative pain, post-operative edema, orbital movement, wound healing, scarring infection, and the post-operative ocular complications such as ectropion, entropion, enophthalmos, scleral show and corneal abrasion.

Postoperative clinical examinations along with radiographic examination was done to evaluate the position of zygoma and determine the adequacy of fracture reduction.

ELIGIBILITY:
Inclusion criteria

* Patients with ZMC fractures that requires open reduction with internal fixation.
* Adult patient between 20 and 50 years with no gender predilections.

Exclusion criteria

* Existing lacerations in the inferior and lateral periorbital regions.
* Comminuted fracture with bone loss.
* Existence of infection at the fracture line.
* Presence of Acute and chronic conjunctival diseases.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
The exposure duration | at the surgery
  The time taken between performing the incision till exposure of the field
postoperative edema | after 1 week
  the postoperative edema was categorized subjectively into mild (just noticeable), mild to moderate (more obvious edema without occlusion of palpebral fissure), moderate to severe (edema partially occluding palpebral fissure), and severe (edema totally occluding palpebral fissure).
change in postoperative pain | 24 hours, 48 hours, 1 week
  assessed through a 10-point Visual Analogue Scale (VAS),(34) (0-1=none,2-4=mild,5-7=moderate,8-10=severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Azarita, Egypt